CLINICAL TRIAL: NCT05752097
Title: Clinical Study of Fibroblast Activating Protein Inhibitor (FAPI) -Mediated 18F Targeted to Evaluate Inflammation and Fibrosis in Renal Diseases
Brief Title: [18F]AlF-NOTA-FAPI-04 PET/CT in Inflammation and Fibrosis in Renal Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SCPHNM
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: 18F-FAPI PET/CT Examination; Renal Puncture Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal inflammatory or fibrotic disease: [18F]AIF-NOTA-FAPI-04 (4.81MBq/Kg) will be injected intravenously according to the patient's body weight. PET/CT examination will be performed 50-60 minutes after the injection of radiotracer. The patients will undergo renal puncture biopsy one day after PET/CT examination.
  Interventions: Device: [18F]AlF-NOTA-FAPI-04 PET/CT examination; Procedure: Renal puncture biopsy

INTERVENTIONS:
Device: [18F]AlF-NOTA-FAPI-04 PET/CT examination — The intravenous radiotracer dose is 1.85-2.59 MBq/kg, and imaging will be performed 50-60 min after radiotracer injection. All patients are required to urinate as much as possible for imaging preparations, which reduces the influence of the residual radiotracer in the renal pelvis and calyces. Some patients with poor renal function (GFR<60 mL/min, urine volume < 1000 mL/24 h) will be given diuretics (Furosemide, 0.57 mg/kg). The scope of the whole-body inspection is from the base of the skull to the base of the thigh, using five to six beds (3 min/bed). The matrix was 128×128, the PET layer thickness was 3 mm, and all PET images are reconstructed iteratively.
Procedure: Renal puncture biopsy — The patients undergo renal puncture biopsy one day after PET/CT examination. Pathological results of renal biopsy will be collected after surgery, including but not limited to: pathological diagnosis, proportion of glomerulosclerosis, extent of inflammatory cell infiltration, and degree of renal interstitial fibrosis.

SUMMARY:
The goal of this observational study is to explore the feasibility of using 18F-labeled FAP molecular probe for PET/CT imaging (18F-FAPI PET/CT) to accurately evaluate inflammation and fibrosis in renal diseases. The main questions it aims to answer are:

* Can 18F-FAPI PET/CT accurately evaluate the inflammation and fibrosis of kidney disease?
* What is the value of 18F-FAPI PET/CT as a non-invasive assessment of inflammation and fibrosis in kidney disease? Participants will receive [18F]AlF-NOTA-FAPI-04 PET/CT and renal aspiration biopsy.

ELIGIBILITY:
Inclusion Criteria:

* The pitients of nephritis or fibrosis disease

Exclusion Criteria:

* Hypertension that is difficult to control with medication, and systolic blood pressure exceeding 160mmHg
* Renal biopsy cannot be performed for severe exclotting disease
* Complicated with chronic liver disease, myocardial infarction, stroke, and malignant tumor
* Unable to cooperate with renal puncture biopsy due to language communication or other problems
* Female patients who are pregnant (or attempting to become pregnant within six months), breastfeeding, or unwilling to use contraception
* Abnormal cardiopulmonary function or mental state, unable to tolerate prone lying for 20 minutes
* Alcohol allergy
* Patients with significant decrease in urine volume due to disease
* Refusal to sign an informed consent form or inability or unwillingness to comply with the investigator-approved protocol
* Other circumstances deemed inappropriate by the investigator for participation in the study.

Ages: 10 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with first clinical diagnosis of nephritis or renal fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value | 30minutes after PET/CT examination
  The extent of renal uptake of FAPI

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Yang X, Liu H, Luo W, Liu H, Lv T, Wang J, Qin J, Ou S, Chen Y. Value of [68Ga]Ga-FAPI-04 imaging in the diagnosis of renal fibrosis. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3493-3501. doi: 10.1007/s00259-021-05343-x. Epub 2021 Apr 7. PMID 33829416
- [Background] Conen P, Pennetta F, Dendl K, Hertel F, Vogg A, Haberkorn U, Giesel FL, Mottaghy FM. [68 Ga]Ga-FAPI uptake correlates with the state of chronic kidney disease. Eur J Nucl Med Mol Imaging. 2022 Aug;49(10):3365-3372. doi: 10.1007/s00259-021-05660-1. Epub 2022 Jan 6. PMID 34988624